CLINICAL TRIAL: NCT02677701
Title: TEACH Trial: Testing the Effect of Adding CHronic Azithromycin to Inhaled Tobramycin. A Randomized, Placebo-controlled, Double-blinded Trial of Azithromycin 500mg Thrice Weekly in Combination With Inhaled Tobramycin
Brief Title: Testing the Effect of Adding Chronic Oral Azithromycin to Inhaled Tobramycin in People With Cystic Fibrosis (CF)
Acronym: TEACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cystic Fibrosis Foundation (Other); CF Therapeutics Development Network Coordinating Center (Network)
Responsible Party: Principal Investigator, David Nichols, MD, Associate Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEACH-IP-15; 1R01HL124053-01A1 (NIH); NICHOL15A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation Therapeutics)
Record Dates: First submitted 2016-01-29; First posted 2016-02-09 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azithromycin (Active Comparator): azithromycin 500mg tablet over-encapsulated to match placebo in appearance, taken by mouth thrice weekly for 6 weeks
  Interventions: Drug: azithromycin; Drug: inhaled tobramycin
- placebo (Placebo Comparator): encapsulated placebo taken by mouth thrice weekly for 6 weeks
  Interventions: Drug: placebo (for azithromycin); Drug: inhaled tobramycin

INTERVENTIONS:
Drug: azithromycin — 500mg tablet over-encapsulated to match placebo
  Other Names: Zithromax
  Arms: azithromycin
Drug: placebo (for azithromycin)
  Arms: placebo
Drug: inhaled tobramycin — clinically prescribed inhaled tobramycin used by subjects participating in the study

SUMMARY:
This is a study to examine the effect of combining chronic oral azithromycin with inhaled tobramycin in adolescent and adult subjects with cystic fibrosis who are chronically infected with P. aeruginosa.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blinded, placebo-controlled trial of azithromycin 500mg taken orally thrice weekly vs. placebo in subjects with cystic fibrosis and chronic airway infection with P. aeruginosa who are utilizing chronic inhaled tobramycin therapy. It will include approximately 120 subjects able to complete a primary 6-week study phase. Subjects will be at least 12 years old with a baseline forced expiratory volume at one second (FEV1) between 25-100% predicted. Subjects will continue to use clinically prescribed inhaled tobramycin cycled on/off every 4 weeks. They will be provided over-encapsulated azithromycin 500mg tablets or placebo during the primary study phase. An optional extension phase will be offered to all subjects completing the primary 6-week study. This 8-week extension phase will include an initial 4 weeks without use of inhaled tobramycin or other inhaled antibiotics, followed by a 4-week period with inhaled tobramycin use. All subjects participating in the extension phase of the study will be provided azithromycin 500mg tablets to be taken thrice weekly for the entire 8-week period.

This study will investigate how use of chronic oral azithromycin affects some of the previously demonstrated benefits to health when using inhaled tobramycin. The primary measurements will focus on lung function. Additional measurements will focus on disease-related quality of life as reported by subjects in the trial. Exploratory outcomes, including measurements of safety, are also planned.

ELIGIBILITY:
Inclusion Criteria:

* 12 years old or older
* documented diagnosis of cystic fibrosis
* written informed consent (and assent when applicable)
* at least two respiratory cultures growing P. aeruginosa within the last 12 months
* FEV1% predicted between 25-100%
* use of at least two cycles of inhaled tobramycin within the last 24 weeks
* Off TISP and other inhaled anti-pseudomonal antibiotics for at least 2 weeks at Visit 1 and remain off of any inhaled antibiotics for an additional 2 weeks before starting inhaled tobramycin
* most recent liver function test results less than 4 times the upper limit of normal, obtained within the last 12 months
* prior or current use of azithromycin for at least four consecutive weeks
* stable clinical status and therapeutic regimen

Exclusion Criteria:

* weight <40 kg
* positive pregnancy test, lactating, or unwillingness to practice a pre-defined form of contraception, which includes abstinence
* inability to perform reproducible spirometry
* inability or unwillingness to cycle off of inhaled tobramycin for one 4-week period and without use of any additional inhaled antibiotics
* respiratory culture with Burkholderia cepacia complex species within 24 months or with nontuberculous mycobacteria within 18 months of screening
* use of intravenous or oral anti-pseudomonal antibiotics within 4 weeks of screening
* use of investigational therapy within 4 weeks of screening
* use of systemic corticosteroids equivalent to a daily dose more than 10mg of prednisone
* use of nelfinavir, warfarin, haloperidol, or methadone (concern of drug interaction with azithromycin)
* initiation of cystic fibrosis transmembrane conductance regulator (CFTR) modulator therapy within 30 days
* ECG abnormality at screening requiring prompt further medical attention, or QTc interval >480 msec for males and >486 msec for females
* any other condition that, in the opinion of the site investigator, would compromise the safety of the subject or quality of the data

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Nichols, MD, Principal Investigator — National Jewish Health
Locations (39):
- United States (39):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital and Health Center at the University of California San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - The Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Maine Medical Partners Pediatric Specialty Care, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Children's Hospital of New York, New York, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center/Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
  - Intermountain Cystic Fibrosis Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: encapsulated placebo taken by mouth thrice weekly for 6 weeks
  placebo (for azithromycin)
  inhaled tobramycin: clinically prescribed inhaled tobramycin used by subjects participating in the study
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 62 | 57
Treated (Participants receiving at least one dose of study drug) | 61 | 54
Completed | 56 | 52
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat population (m-ITT) defined as all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 61 | 54 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (9.9) | 26.5 (9.7) | 26.3 (9.8)
Age, Customized [Count of Participants; unit: Participants]
  Age Distribution: ≥ 12 to < 18 years | 14 | 12 | 26
  Age Distribution: ≥ 18 to < 30 years | 28 | 25 | 53
  Age Distribution: ≥ 30 years | 19 | 17 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 32 | 28 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 52 | 47 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 55 | 49 | 104
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 61 | 54 | 115
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants] — Other refers to participants with either two known, non-F508 del CF mutations, or one known, non-F508 del CF mutation and one unidentified allele which has not been classified as a CF mutation. Unidentified refers to participants with 2 alleles that have not been classified as CF mutations.
  Participants
    Delta F508 Homozygous | 38 | 35 | 73
    Delta F508 Heterozygous | 17 | 11 | 28
    Other | 6 | 7 | 13
    Unidentified | 0 | 0 | 0
    Not Available | 0 | 1 | 1
FEV1 [Mean (Standard Deviation); unit: liters] — FEV1 is the forced expiratory volume in one second.
  liters | 2.59 (0.81) | 2.50 (0.85) | 2.55 (0.83)
ppFEV1 Category [Count of Participants; unit: Participants] — FEV1 percent of predicted (ppFEV1) is calculated using the Global Lung Initiative multi-ethnic reference equations for ages 3-95.
  Participants
    ≥ 25% to < 50% | 11 | 11 | 22
    ≥ 50% to < 75% | 22 | 16 | 38
    ≥ 75% | 28 | 27 | 55
Current Tobramycin Formulation [Count of Participants; unit: Participants]
  Tobramycin Inhaled Solution | 33 | 28 | 61
  Tobramycin Inhaled Powder | 28 | 26 | 54
History of Azithromycin Use at Baseline [Count of Participants; unit: Participants] — Current use is defined as use of chronic oral azithromycin for the past 30 days (can be either 3x/week or daily dosing).
  Participants
    Current User | 51 | 43 | 94
    Non-Current User | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in Lung Function
Description: Relative change in FEV1 volume (L) from enrollment at week 0 to the end of the 4-week period with inhaled tobramycin at week 6
Time Frame: baseline (week 0) to week 6 (6 week period)
Population: Participants in the m-ITT population with spirometry measurements of FEV1 liters at both baseline (week 0) and week 6.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 56 | 52
percent change | 1.69 (10.39) | -1.95 (10.73)
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.0846, Regression, Linear; Adjusted for baseline: ppFEV1 (25%-50%, >50%-75%, >75%), azithromycin use (current vs. non-current), inhaled tobramycin type (powder vs. solution); Mean Difference (Net) = 3.44, 95% CI 2-sided [-0.48 to 7.35]

2. Secondary Outcome: Relative Change in Lung Function
Description: Relative change in FEV1 (L) from the beginning of the 4-week period with inhaled tobramycin at week 2 to the end of the 4-week period with inhaled tobramycin at week 6
Time Frame: week 2 to week 6 (4 week period)
Population: Participants in the m-ITT population with spirometry measurements of FEV1 liters at both week 2 and week 6.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 56 | 52
percent change | 0.44 (8.86) | -0.91 (11.41)
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.51, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.31, 95% CI 2-sided [-2.64 to 5.26]

3. Secondary Outcome: Change in Cystic Fibrosis Respiratory Symptom Diary - Chronic Respiratory Infection Symptom Score (CFRSD-CRISS)
Description: Absolute change in CFRSD-CRISS from enrollment at week 0 to the end of the 4-week period with inhaled tobramycin at week 6. The Cystic Fibrosis Respiratory Symptoms Diary asks a participant to state the extent of 8 respiratory symptoms: difficulty breathing, feverishness, tiredness, chills or sweats, coughing, coughing up mucus, tightness in the chest, and wheezing. Each respiratory symptom is assigned a score from 0-4 based on the response, with zero corresponding to the absence of the symptom and four corresponding to symptom being present "a great deal" or "extremely." A summed score (ranging from 0-24) is calculated for each participant and converted to a final score with a range of 0 to 100, where lower scores indicate improvement of symptoms.
Time Frame: baseline (week 0) to week 6 (6 week period)
Population: Participants in the m-ITT population with CFRSD-CRISS diaries at both baseline (week 0) and week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 56 | 52
score on a scale | -2.3 (11.4) | 0.6 (9.8)
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.17, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -2.89, 95% CI 2-sided [-7.01 to 1.22]

4. Secondary Outcome: Change in Cystic Fibrosis Questionnaire - Revised Respiratory Symptom Score (CFQ-R RSS)
Description: Absolute change in the CFQ-R RSS from enrollment at week 0 to the end of the 4-week period with inhaled tobramycin at week 6. Age appropriate versions of Cystic Fibrosis Questionnaire - Revised ask a participant from 4 to 6 questions related to respiratory symptoms. The Respiratory Domain Scaled Score is calculated as follows: 100*[sum of {responses-1}] / [{number of responses}*3] only if [number of responses] ≥ [number of possible responses]/2; otherwise the score is set to missing. The scaled score ranges from 0 to 100 and higher scores indicate improvement of symptoms.
Time Frame: baseline (week 0) to week 6 (6 week period)
Population: Participants in the m-ITT population with CFQ-R respiratory symptom scores at both baseline (week 0) and week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 53 | 52
score on a scale | 1.0 (14.0) | -0.5 (12.5)
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.56, Regression, Linear — Adjusted for baseline: ppFEV1 (25%-50%, >50%-75%, >75%), azithromycin use (current vs. non-current), inhaled tobramycin type (powder vs. solution); Mean Difference (Net) = 1.53, 95% CI 2-sided [-3.70 to 6.77]

5. Other Pre Specified Outcome: Change in Sputum Pseudomonas Aeruginosa Bacterial Density
Description: Absolute change in log10 transformed quantitative Pseudomonas aeruginosa (Pa) bacterial density as measured by colony forming units (CFUs) per mL of sputum from enrollment at week 0 to the end of the 4-week period with inhaled tobramycin at week 6. Culture results below the lower limit of detection of 1x10^2 were set to 1/2 of that LLD prior to log transformation.
Time Frame: baseline (week 0) to week 6 (6 week period)
Population: Participants in the m-ITT population with Pseudomonas aeruginosa sputum culture results at both baseline (week 0) and week 6.
Measure: Mean (Standard Deviation); unit: log10(CFUs/mL)
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 29 | 35
log10(CFUs/mL) | 0.3 (1.7) | -0.5 (1.2)
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Test type: Superiority; p = 0.043, Regression, Linear — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = 0.75, 95% CI 2-sided [0.03 to 1.47]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/54
Serious Adverse Events (participants affected / at risk) | 4/61 | 3/54
Other Adverse Events (participants affected / at risk) | 22/61 | 32/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=61) | Placebo (N=54)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=61) | Placebo (N=54)
Headache (Nervous system disorders) | 8 (15) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 16 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (8)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT02677701/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02677701/SAP_001.pdf